CLINICAL TRIAL: NCT04164706
Title: Quality of Recovery and Perioperative Hypothermia in Elective Colectomy Patients: A Feasibility Study of a Blinded Randomised Controlled Trial
Brief Title: HEAT HumiGard Evaluation Study
Acronym: HEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Principal Investigator, Judith White, Trial Manager, Cardiff and Vale University Health Board
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19/MAR/7616
Record Dates: First submitted 2019-10-30; First posted 2019-11-15 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Laparoscopic Colorectal Surgery
Keywords: Colorectal Cancer; Colorectal Surgery; Laparoscopic; Hypothermia
MeSH Terms: conditions — Colorectal Neoplasms; Hypothermia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Feasibility study - 40 patients to be randomised 1:1 to two groups - 50% receiving HumiGard and 50% receiving standard care alone
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Everyone will be blinded except for one member of the theatre staff who will operate the HumiGard, and the research team member who performs the randomisation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HumiGard (plus standard care) (Experimental): HumiGard device will be used to provide warmed humidified CO2 for insufflation during laparoscopic surgery. The device will be used alongside standard methods of keeping the patient warm in theatre. The theatre team will monitor the patient's temperature at regular time points before, during and after surgery. Warmed fluids, forced air warming devices or warmed blankets will be used as required to maintain normothermia.
  Interventions: Device: HumiGard device
- Standard Care (with sham HumiGard device). (Sham Comparator): Patients will receive standard methods of keeping the patient warm in theatre. The theatre team will monitor the patient's temperature at regular time points before, during and after surgery. Warmed fluids, forced air warming devices or warmed blankets will be used as required to maintain normothermia.
  A sham HumiGard device will be used in the standard care arm. This will be the same HumiGard device as is in the intervention arm. However, the sham device will be turned "off" so that the gas delivered to the peritoneal cavity for insufflation is not heated or humidified. The sham device will deliver CO2 (as is the case for current standard practice in the hospital) through the HumiGard tubing. The sham device will look and sound the same as the active intervention arm where the HumiGard device is switched "on" and is delivering warm, humidified CO2 to the peritoneal cavity.
  Interventions: Other: Standard care (with sham HumiGard device)

INTERVENTIONS:
Device: HumiGard device — HumiGard is a CE marked device that delivers warmed humidified CO2 during laparoscopic surgery
  Other Names: HumiGard Surgical Humidification System SH870
  Arms: HumiGard (plus standard care)
Other: Standard care (with sham HumiGard device) — Standard methods of keeping the patient warm whilst in theatre, including warmed IV fluids, warming blankets/forced air warming devices.
  Arms: Standard Care (with sham HumiGard device).

SUMMARY:
During long surgical procedures under general anaesthetic, patients' body temperatures sometimes drop below 36°C. This is classified as hypothermia. These low temperatures are associated with medical complications and surgical wound infections. Despite various warming methods used during surgery a significant number of patients experience hypothermia during surgery. During laparoscopic procedures, standard practice is to use dry, unwarmed carbon dioxide (CO2) to inflate the peritoneum (insufflation). This may contribute to the risk of hypothermia and cause tissue desiccation.

HumiGard is a CE marked device which humidifies and heats CO2 for insufflation. It is used together with other standard methods of keeping patients warm. Other studies suggest that the HumiGard device may prevent hypothermia, and help patients recover more quickly and with fewer problems after surgery.

The investigators aim to find out whether the HumiGard device used with standard practice, gives better outcomes for patients, compared to standard care alone. To do this, the investigators first need to work out if such a study would be feasible to do and therefore whether a larger study can be done.

A total of 40 patients who are having a laparoscopic colectomy operation (where a portion of their bowel is removed) will be recruited. Half will be treated with the HumiGard device plus standard care and half will be treated with a sham HumiGard device plus standard care. Patients will be allocated to one of these groups by random chance. Neither the patient, the surgeon, nor the assessor will know which treatment the patient is having.

The investigators will measure patients' temperature during surgery, and also patients will be asked to complete a validated questionnaire to measure their quality of recovery and pain following surgery. The feasibility study will aim to highlight the most appropriate outcomes to be measured in a larger RCT.

DETAILED DESCRIPTION:
Laparoscopic surgery involves filling the peritoneal cavity with carbon dioxide (CO2) gas (insufflation) to increase the working and viewing space in the abdomen. It is standard care in the United Kingdom (UK) to use dry, unwarmed CO2. There is evidence that dry, unwarmed insufflation is associated with tissue desiccation and intraoperative hypothermia showing that insufflation of cool dry gas resulted in a temperature drop of 1.3-1.7°C. Despite active warming methods, perioperative hypothermia is common. One study demonstrated that nearly half of patients had continuous core temperatures of 36°C for more than an hour.

HumiGard (Fisher and Paykel Healthcare) is a CE marked medical device designed to humidify and heat CO2 for insufflation. A meta-analysis included 13 studies (total of 796 patients) comparing warmed, humidified CO2 insufflation compared to unwarmed, dry CO2 in patients having a range of procedures. There was a significant difference in mean core temperature change, and an effect size of +0.3°C (95% confidence interval [CI]: 0.1-0.6). This was more pronounced in studies of long procedures (80 min). Another meta-analysis of 15 studies (1026 patients) demonstrated a small beneficial effect on immediate post-operative pain but not at day 1 or 2. Warmed, humidified CO2 reduced the risk of intraoperative hypothermia (p=0.004) but postoperative core temperatures were not significantly different (10 studies, 718 patients). No differences were observed in analgesic consumption, length of stay, or procedure duration.

This is a blinded, randomised controlled feasibility study on 40 patients receiving laparoscopic colorectal resectional surgery at a single site (University Hospital of Wales) and treated with either the HumiGard device plus standard care (20 patients) or a sham HumiGard device plus standard care (20 patients).

This study will assess various aspects of a proposed larger pragmatic blinded, RCT evaluating whether HumiGard insufflation device, when used with standard care, can improve patients' quality of recovery after laparoscopic colectomy surgery.

The feasibility study will aim to highlight the most appropriate outcomes to be measured in a main RCT, particularly looking at the role of Quality of Recovery (QoR-40) questionnaire or continuous temperature measurements. The investigators will assess whether the outcomes of the study are suitable, achievable and measurable. The study will assess recruitment, ability to blind operating surgeon with a sham HumiGard device, use of urinary temperature probe compared to standard temperature monitoring in theatre, use of QoR-40 and visual analogue score (VAS) pain score by patients preoperatively (for a baseline score) and on post-operative day (POD) 1, 3 and 30, analgesia use, and intraoperative patient warming techniques. Length of stay in hospital from procedure to discharge (or until medically fit for discharge) will also be recorded and reported.

Furthermore, methods for analysing the postoperative complication rate will be evaluated. Complications will be recorded at POD1, POD3, upon discharge and POD30. Their severity will be graded using the Clavien-Dindo scale, a widely used and valid method for grading severity of surgical complications which helps to reduce subjectivity. The Comprehensive Complication Index (CCI) will then be used to create a composite score (0-100) for each patient.

ELIGIBILITY:
The study will recruit patients undergoing an elective laparoscopic colorectal resection operation for any pathology. The patients will be over 18, and able to provide informed consent.

Inclusion Criteria:

* ≥18 years of age
* Participant is willing and able to give informed consent
* Scheduled for elective laparoscopic, segmental or total colectomy

Exclusion Criteria:

* Unable to complete study documentation
* Lack of capacity or not willing to give consent
* Open procedure planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
To assess if a recruitment rate of at least 6 patients per month in a tertiary centre is achievable and identify any barriers to recruitment | Post-operative day 1
  The recruitment rate will be assessed using the "screening and recruitment log" which will record the number of patients recruited each month and reasons for non-recruitment will be described.

SECONDARY OUTCOMES:
Number of patients who complete the QoR-40 questionnaire and VAS score | Pre-operatively and post-operative days 1,3,30
  The number of patients who successfully complete the QoR-40 questionnaire and VAS score pre-operatively and at post-operative days 1,3,30 will be measured.
Number of patients who have successful continuous intra-operative temperature readings using a urinary temperature probe | Intra-operatively
  The number of patients who have successful continuous intra-operative temperature readings using a urinary temperature probe will be measured. The feasibility of using these data to identify periods of intraoperative hypothermia will also be assessed.
Number of cases in which the treating surgeon correctly predicted the study arm allocation of the patient (HumiGard vs sham device). | Intra-operatively
  The number of cases in which the treating surgeon correctly predicted the study arm allocation of the patient (HumiGard vs sham device) will be recorded in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Reeves, MD, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- Dept of Surgery, Cardiff & Vale University Health Board, Cardiff, United Kingdom